CLINICAL TRIAL: NCT06068725
Title: T The Effect Of Video Training On Symptom Management And Quality Of Life In Patients Over 65 Years Of Age Wıth Heart Failure
Brief Title: The Effect of Video Training o Symptom Management With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Pinar YEL, Lecturer, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EU-NF-PY-01
Record Dates: First submitted 2023-09-29; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure
Keywords: Quality of Life; Geriatrics; Nursing
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: It consists of two groups, application and control, and three follow-ups.
Who Masked: Participant, Outcomes Assessor
Masking Description: In the study, groups were determined by block randomization. The randomization list was created by block randomization according to New York Heart Association (NYHA) classification.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No invention: Control Group (No Intervention): Data collection tools were applied to individuals in the control group on day 0 (Z0), day 30 (Z1) and day 90 (Z2) of follow-up. Data collection tools applied to the control group are as follows: Patient Introduction Form, Heart Failure Symptom Status Scale, Minnesota Living with Heart Failure Questionnaire,Michel Uncertainty in Illness Scale - Community Form.
- Experimental: application group (Experimental): Two 15-minute training videos (30 minutes in total) prepared for symptom management will be shared on the phones of the patients/relatives in the application group and the patients and their relatives will be informed by watching the training video.Data collection tools were applied to individuals in the application group on day 0 (Z0), day 30 (Z1) and day 90 (Z2) of follow-up. Data collection tools applied to the application group are as follows: Patient Introduction Form, Heart Failure Symptom Status Scale, Minnesota Living with Heart Failure Questionnaire,Michel Uncertainty in Illness Scale - Community Form.
  Interventions: Behavioral: Training videos

INTERVENTIONS:
Behavioral: Training videos — After determining the application and control groups in the research, the purpose of the research was explained to both groups. The mobile phone usage skills of the individuals who will be included in the application group were evaluated with the Digital Literacy Scale. Training videos for 15 people each (30 minutes in total) regarding symptom management were shared on the phones of the patients/relatives in the application groups, and the patients and their relatives were informed and watched the training video. Data collection forms would be filled out before the application (Z0), on the 30th day of the application (Z1), and on the 90th day of the application (Z2).
  Arms: Experimental: application group

SUMMARY:
The purpose of this clinical study is to compare the effect of video-assisted training on the quality of life and symptom management of patients over the age of 65. The main questions it aims to answer are:

-Is there a difference between symptom management and quality of life between the first and last follow-up periods of patients in the application and control groups?

DETAILED DESCRIPTION:
Heart failure is the primary disease of old age. 20% of the reasons for hospital admission for patients aged 65 and over are due to heart failure.The most common symptoms in patients with heart failure are; fatigue, weakness, dyspnea, orthopnea, paroxysmal nocturnal dyspnea, edema and changes in mental status.Due to these physical symptoms; there is a decrease in the functional capacity of patients, difficulty in performing daily life activities, inability to perform self-care, and the incidence of depression and anxiety increases.

In symptom management of patients with heart failure; these include knowing the clinical course of the disease, adapting to the disease and treatment, monitoring symptoms, educating the patient on self-care, and regular follow-up after discharge.It is stated that with patient education given to individuals in a planned and regular manner, the frequency and severity of the symptoms experienced decreases, the management and control of the disease is ensured, and thus the patient's quality of life is increased by creating the necessary behavioral changes.Due to the increase in the number of internet users in patient education, web-based education becomes more prominent.Thanks to video training, patients will be able to experience a permanent learning process by accessing the training content wherever they want, as often as they want.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and above
* Volunteer to participate in the research
* Diagnosed with heart failure at least six months ago
* He/she/his relative has internet access and can use a smartphone
* Digital literacy scale score over 17
* Class I, II, III according to NYHA classification

Exclusion Criteria:

* Under 65 years of age
* Known serious vision and hearing problems
* With cognitive impairment

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Heart Failure Symptom Status Scale | Three months
  It measures the presence, frequency and severity of seven basic symptoms, such as dyspnea during the day, dyspnea when lying down, fatigue, chest pain, edema, sleep problems, dizziness or dizziness, which are the most common in heart failure patients, and the degree to which each of these symptoms affects the patient.When the patient expresses the "zero" option, this indicates that the patient does not have the relevant symptom. To calculate each symptom, all values given by patients for frequency, severity and discomfort are added together. The scores that can be obtained from the scale vary between 0-84.

SECONDARY OUTCOMES:
Minnesota Living with Heart Failure Questionnaire | Three months
  Disease-specific heart failure and its treatment in patients' lives; It evaluates its effects and perceptions in physical, socio-economic and psychological dimensions.The total score on the scale varies between 0-105. A low score on the scale indicates a high quality of life
Michel Uncertainty in Illness Scale - Society Form | Three months
  The scale reveals the uncertainty experienced by individuals with chronic diseases during periods when they are not hospitalized. The Turkish version of the scale consists of 20 items. The scale is evaluated through three sub-dimensions and a total score: "perception of the current situation", "perception of understanding" and "uncertainty".The score that can be obtained from the scale varies between 20 and 100, with the average being 60. An increase in the score obtained from the scale is interpreted as an increase in disease uncertainty.

CONTACTS AND LOCATIONS:
Overall Officials: Pinar YEL, Principal Investigator — Ege University
Locations (2):
- Turkey (Türkiye) (2):
  - Dr. Sadi Konuk Training and Research Hospita, Istanbul
  - Istanbul Yeni Yüzyıl University Private Gaziosmanpaşa Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No